CLINICAL TRIAL: NCT04424901
Title: A Randomized, Open-label Study of the Vascular and Microbiologic Efficacy of Dipyridamole Plus Standard Care vs. Standard Care in Hospitalized COVID19 Patients
Brief Title: Trial of Open Label Dipyridamole- In Hospitalized Patients With COVID-19
Acronym: TOLD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: reduction of Hospitalized COVID patients at UConnHealth
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Bruce Liang, Professor of Medicine School of Medicine, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-192-2.F
Record Dates: First submitted 2020-05-29; First posted 2020-06-11 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Pneumonia; Vascular Complications
MeSH Terms: interventions — Dipyridamole

STUDY DESIGN:
Intervention Model Description: Randomized Open Label Study Standard Care vs. Standard Care with Dipyridamole
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Care (Placebo Comparator): Hospitalized patients meeting screen criteria receive standard Hospital care from which clinical event and lab data are collected.
  Day 3,6 & 9 research samples will be used for obtaining immunological profiles as well as metabolomic profiling and whole genome sequencing for discovery of new biomarkers/ genomic regions that confer increased susceptibility to infection and DIP treatment efficacy or safety. Other samples will be obtained for microbiome and viral analyses.
  Data collection ends on day 9.
  Interventions: Drug: Placebo
- Standard Care with Dipyridamole (Experimental): For this arm, Dipyridamole 100 mg, tid is given for 7 days. Hospitalized patients meeting screen criteria receive standard Hospital care from which clinical event and lab data are collected.
  Day 3,6 & 9 research samples will be used for obtaining immunological profiles as well as metabolomic profiling and whole genome sequencing for discovery of new biomarkers/ genomic regions that confer increased susceptibility to infection and DIP treatment efficacy or safety. Other samples will be obtained for microbiome and viral analyses.
  Data collection ends on day 9.
  Interventions: Drug: Dipyridamole Tablets

INTERVENTIONS:
Drug: Placebo — Daily dose while hospitalized up to 9 days
  Arms: Standard Care
Drug: Dipyridamole Tablets — Daily dose while hospitalized up to 9 days
  Other Names: Persantine
  Arms: Standard Care with Dipyridamole

SUMMARY:
Brief Summary:

The goal here is to evaluate dipyridamole in treating respiratory tract infection and circulatory dysfunction due to SARS-CoV-2 coronavirus in hospitalized CVID-19 patients.

Infection with SARS-CoV-2 causes human COVID-19 (HCoV-19). The infection is associated with a deleterious inflammatory response and a prothrombotic state in addition to tissue damage from direct viral entry and proliferation. Dipyridamole has anti-platelet and anti-inflammatory effects. The drug was recently demonstrated to have anti-SARS-Cov-2 effect primarily in vitro. The concentration causing anti-viral effect in vitro is within that in the blood of humans taking this drug. As an oral tablet, it has the advantage of easy administration.

Anti thrombotic, anti viral and anti inflammatory actions of this drug may be efficacious and safe in hospitalized subjects

DETAILED DESCRIPTION:
The original protocol stipulated an enrollment of 100 patients, randomized in a 1 to 1 distribution of treatment versus control [placebo] group. However, the study was terminated because of insufficient enrollment due to the dramatic reduction in the number of hospitalized COVID patients.

A total of 41 patients were randomized prior to study termination. Detailed reports and overall results were reviewed for all patients.

Adverse event occurrences were similar in groups. Given the severity of COVID, these numbers were not unexpected.

The DSMC concluded that all the AEs seen in study subjects are either unrelated or probably unrelated to the TOLD study intervention.

The DSMC reviewed the primary outcome results. No statistically significant change in either the platelet count or the D-dimer results.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age.
2. COVID-19 positive by PCR and hospitalized for respiratory infection with a range of respiratory severity as follows.

   Moderate ● Diagnosed with SARS-CoV-2 infection by standard RT-PCR assay or equivalent testing

   ● Symptoms of moderate illness with COVID-19, which could include:

   o Fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms; shortness of breath with exertion
   * Clinical signs suggestive of moderate illness with COVID-19, such as:

     o RR ≥ 20, HR ≥ 90, SaO2 ≥93% on room air or requires ≤2L oxygen by nasal cannula (NC) in order maintain SaO2 ≥93%, fever >38.3 Celsius
   * No clinical signs indicative of Severe or Critical Illness Severity

   Severe
   * Diagnosed with SARS-CoV-2 infection by standard RT-PCR assay or equivalent testing
   * Symptoms suggestive of severe systemic illness with COVID-19, which could include:

     o any symptom of Moderate Illness; shortness of breath at rest or respiratory distress
   * Clinical signs indicative of severe systemic illness with COVID-19, such as

     o RR ≥ 30, HR ≥ 125, requires > 2L oxygen by NC in order maintain SaO2 ≥93%, PaO2/FiO2 <300
   * No criteria for Critical Severity

   Critical ● Diagnosed with SARS-CoV-2 infection by standard RT-PCR assay or equivalent testing
   * Evidence of critical illness, defined by at least 1 of the following:

     * Respiratory failure defined based on resource utilization requiring at least 1 of the following:

       ◙, Oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20L/min with fraction of delivered oxygen ≥0.5), noninvasive positive pressure ventilation, ECMO, or clinical diagnosis of respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation)
     * Shock (defined by SBP < 90 mm Hg, or Diastolic BP < 60 mm Hg or requiring vasopressors)
     * Multiple organ dysfunction/failure
3. Able to give written informed consent in English to participate in the study by patient.

   -

Exclusion Criteria:

* Exclusion Criteria:

  1. Inability to swallow or ingest oral medication in either tablet form or in suspension form.
  2. Patient is known to be pregnant
  3. Patients with a history of allergy or hypersensitivity to dipyridamole
  4. Patient is unable to consent -intubated, on mechanical ventilation
  5. Bleeding disorders (e.g. thrombocytopenia with platelet counts < 50,000)
  6. Existing severe medical illnesses unrelated to Covid-19 infection such as end stage heart, kidney, liver disorders;

     or hepatic insufficiency defined as liver enzymes ≥5 times upper limit normal if baseline is normal or 5 times baseline if baseline is abnormal.

     Metastatic cancer as well as those with severe coronary artery disease, unstable angina, STEMI, NSTEMI, hypotension (systolic blood pressure <90mmHg), myocarditis, bradycardia with resting heart rate less than 60 bpm, atrioventricular block without pacemaker.

     Those with myasthenia gravis and those treated with cholinesterase inhibitors
  7. Patient is enrolled in a clinical trial for another investigational drug designed to test for efficacy for SARS-CoV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-05-03 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Liang, MD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from Acute Care University Hospital Units May 2020 to March 2022
Pre-assignment Details: At Consent, subjects are randomized to Placebo or Dipyridamole group.
Groups:
- Standard Care With Dipyridamole: For this arm, Dipyridamole 100 mg, tid is given for 7 days. Hospitalized patients meeting screen criteria receive standard Hospital care from which clinical event and lab data are collected.
  Day 3,6 & 9 research samples will be used for obtaining immunological profiles as well as metabolomic profiling and whole genome sequencing for discovery of new biomarkers/ genomic regions that confer increased susceptibility to infection and DIP treatment efficacy or safety. Other samples will be obtained for microbiome and viral analyses.
  Data collection ends on day 9.
  Dipyridamole: Dipyridamole-100mg taken 3 times a day by mouth for 7 days.
Period: Overall Study
Arm/Group | Standard Care | Standard Care With Dipyridamole
Started | 21 | 20
Completed | 4 | 4
Not Completed | 17 | 16
Not completed — patients were discharged prior to Hospital Day 9 | 17 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Standard Care With Dipyridamole | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.62 (14.06) | 60.75 (13.89) | 60.17 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 15 | 10 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 18 | 12 | 30
  Race: Asian | 1 | 0 | 1
  Race: Black/African American | 1 | 4 | 5
  Race: Hispanic/Latino | 1 | 3 | 4
  Race: Not Reported | 0 | 1 | 1
COVID-19 -moderate or severe [Count of Participants; unit: Participants] | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: D-dimer
Description: Percent Change from Baseline [Day Zero] to last study measure (Day 3, Day 6 or Day 9)
Time Frame: up to 9 days
Population: Percent Change from Baseline
Measure: Median (Inter-Quartile Range); unit: Percent Change of D-Dimer (ng/mL)
Arm/Group | Standard Care | Standard Care With Dipyridamole
Number analyzed (Participants) | 17 | 16
Percent Change of D-Dimer (ng/mL) | 2.99 [-17.12 to 85.63] | -10.09 [-22.06 to 6.08]

2. Primary Outcome: Platelet Count
Description: Percent Change from Baseline [Day Zero] to last study measure (Day 3, Day 6 or Day 9)
Time Frame: up to 9 days
Population: Percent Change (%) from Baseline
Measure: Mean (Standard Deviation); unit: Percent Change of 10^3 Platelets/uL
Arm/Group | Standard Care | Standard Care With Dipyridamole
Number analyzed (Participants) | 17 | 15
Percent Change of 10^3 Platelets/uL | 27.45 (34.94) | 35.48 (37.52)

3. Secondary Outcome: Viral Detection
Description: Evaluate for a non-detection from nasopharyngeal swab and in stool
Time Frame: 9 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Survival
Description: Survival Status Alive
Time Frame: 9 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Inflammatory Markers
Description: Change in the markers CRP/Ferritin
Time Frame: 9 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Blood Markers
Description: Change in Lymphocyte Count/ Fibrinogen/Cardiac Troponin
Time Frame: 9 days
Reporting Status: Not Posted

7. Other Pre Specified Outcome: PT PTT
Description: Coagulation System
Time Frame: 9 days
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Pulmonary Status
Description: Change in SpO2/ imaging
Time Frame: 9 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Clinical Status
Description: Change in fever, cough, sputum
Time Frame: 9 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Mortality assessed up to 30 days beyond date of enrollment
Arm/Group | Standard Care | Standard Care With Dipyridamole
All-Cause Mortality (participants affected / at risk) | 2/21 | 2/20
Serious Adverse Events (participants affected / at risk) | 5/21 | 7/20
Other Adverse Events (participants affected / at risk) | 9/21 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=21) | Standard Care With Dipyridamole (N=20)
Death NOS (General disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Alanine Aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=21) | Standard Care With Dipyridamole (N=20)
Headache (Nervous system disorders) | 5 (5) | 4 (4)
Fever (General disorders) | 4 (4) | 4 (4)
Increase Alanine Aminotransferase (Investigations) | 2 (2) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Increase Aspartate Aminotransferase (Investigations) | 1 (1) | 4 (4)
Hypotension (Vascular disorders) | 2 (2) | 4 (4)
Pain (General disorders) | 4 (4) | 3 (3)
Hypertension (Vascular disorders) | 4 (4) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 3 (3) | 3 (6)
Sinus Bradycardia (Cardiac disorders) | 4 (4) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Platelet Count decreased (Investigations) | 1 (1) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
No data obtained beyond 9 days of enrollment. If discharged from care, phone follow up limited to data provided by subject report, up to day 9.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT04424901/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT04424901/ICF_001.pdf